CLINICAL TRIAL: NCT05521113
Title: Feasibility of Home-based Pulmonary Rehabilitation With Remote Monitoring in Pulmonary Arterial Hypertension
Brief Title: Home-based Pulmonary Rehabilitation With Remote Monitoring in Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hilary M. DuBrock, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 22-000414
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home Rehabilitation Monitoring System: Subjects will complete a home pulmonary rehabilitation program while using a home rehabilitation monitoring system and completing health coaching calls.
  Interventions: Behavioral: Home Rehabilitation Monitoring System; Behavioral: Health coaching calls

INTERVENTIONS:
Behavioral: Home Rehabilitation Monitoring System — The system consists of a small activity monitor worn on the wrist and a pulse oximeter worn on the finger while exercising. Simple exercises will be completed daily and the monitors will send information to a rehabilitation coach during a 12-week period.
Behavioral: Health coaching calls — 12 telephone-based health coaching calls over a 12-week period

SUMMARY:
The purpose of this study is to test new technology and health coaching aimed to help people with PAH become more physically active in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH, confirmed by right heart catheterization (mean pulmonary artery pressure of 20 mmHg or greater, pulmonary vascular resistance of 3.0 Woods units or greater, Pulmonary capillary wedge pressure of 15 mmHg or lower).
* On PAH-specific therapy which is at stable dosing (i.e., not currently titrating therapy).
* NYHA class II-III symptoms.
* Able to complete a six-minute walk test.

Exclusion Criteria:

* Patients experiencing syncope or exertional syncope.
* Patients not experiencing exertional dyspnea.
* Inability to walk.
* Patients currently in pulmonary rehab or having completed pulmonary rehab within three months (unlikely to improve).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified with the medical diagnoses of Pulmonary Arterial Hypertension (PAH) from the Mayo Clinic in Rochester, MN PH clinic.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 weeks
  Number of adverse events attributed to home-based pulmonary rehabilitation

SECONDARY OUTCOMES:
Change in EmPHasis-10 Quality of Life Survey | Baseline, 3 months
  Measured using the EmPHasis-10 to determine how pulmonary hypertension affect subject's life. 10-item self-reported questionnaire, total score 0-50 with higher scores indicating worse outcomes or quality of life.
Change in PAH-SYMPACT domain scores Quality of Life | Baseline, 3 months
  Measured using the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire to assess pulmonary arterial hypertension symptoms over the past 24 hours and 7 days. 23-item self-reported questionnaire, total score 0-89 with higher scores indicating worse outcomes or quality of life.
Change in self-management abilities | Baseline, 3 months
  Measured by the Self-Management Ability Scale (SMAS-30) to determine self-management abilities. 30-item self-reported questionnaire, average overall scores 5-30 with higher scores indicating higher self-management abilities.
Change in daily physical activity | Baseline, 3 months
  Number of daily steps captured by the Home Rehabilitation Monitoring System
Change in exercise capacity | Baseline, 3 months
  Measured by 6-minute walk exercise captured by the Home Rehabilitation Monitoring System

CONTACTS AND LOCATIONS:
Overall Officials: Hilary DuBrock, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials